CLINICAL TRIAL: NCT04380571
Title: Biofeedback Versus Bilateral Transcutaneous Electrical Nerve Stimulation in the Treatment of Functional Non-retentive Fecal Incontinence
Brief Title: Biofeedback Vs Electrical Stimulation in Treatment of Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olfat Ibrahim Ali, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fecal incontinence
Record Dates: First submitted 2020-04-29; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Fecal Incontinence; Encopresis; Fecal Soiling
Keywords: Fecal incontinence; Biofeedback; Transcutaneous posterior tibial nerve stimulation; Childern
MeSH Terms: conditions — Fecal Incontinence; Encopresis | interventions — Biofeedback, Psychology; Electric Stimulation; Exercise

STUDY DESIGN:
Intervention Model Description: The current prospective randomized controlled study included 93 children with FNRFI who were randomly divided and allocated into 3 groups. were managed by conventional methods through Kegal exercises and dietetic regulation where they had received bulky food including vegetables, fruits bran and cereals. Fast foods, spicy drinks and caffeine should be limited in child's diet. Local hygiene and zinc oxide application to the perianal skin were advised to prevent skin excoriation.Biofeedback group treated by biofeedback therapy in addition to traditional treatment, while the third group is the electrical stimulation group received bilateral (TPTNS) in addition to the traditional treatment. Initial manometric findings including resting pressure (mm hg), squeeze pressure (mm hg), 1st sensation (cm water), 1st urge (cm water), and intense urge (cm water) were recorded and repeated after 3 and 6 months together with incontinence score recorded in using St' Mark's (Varizey).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biofeedback (Experimental): Biofeedback therapy in addition to the conventional measures done in the control Group. It was performed in the same position used for baseline manometry. The used protocol included strength and sensory training, twice weekly for 3 months. Strength training was performed by a double-lumen rectal PVC balloon clothed catheter (MMS U-72210).
  Interventions: Device: Biofeedback
- Electrical Stimulation (Experimental): Bilateral (TPTNS); was applied with an electrode above the medial malleolus A second electrode) was applied just below the same malleolus. Electrical stimulation with a low-frequency current (10 Hz), and adjustable intensity. The procedure was done for 20-30 minutes, three times per week for 3 months together with the conventional maneuvers applied in the control group.
  Interventions: Device: Electrical stimulation
- Control group (Active Comparator): were managed by conventional methods through Kegal exercises and dietetic regulation where they had received bulky food including vegetables, fruits bran and cereals. Fast foods, spicy drinks and caffeine should be limited in child's diet. Local hygiene and zinc oxide application to the perianal skin were advised to prevent skin excoriation.
  Interventions: Other: Traditional treatment

INTERVENTIONS:
Device: Biofeedback — Biofeedback therapy in addition to the conventional measures done in the control Group. It was performed in the same position used for baseline manometry. The used protocol included strength and sensory training, twice weekly for 3 months. Strength training was performed by a double-lumen rectal PVC balloon clothed catheter (MMS U-72210).
  Arms: Biofeedback
Device: Electrical stimulation — A positive auto adhesive electrode was applied above the medial malleolus over the S3 dermatome. A second negative electrode was applied just below the same malleolus. Both electrodes were linked to an electrical stimulation device ( EMS physio Ltd, OX129 F, England) with a low frequency current (10 Hz), and adjustable intensity.
  Other Names: Posterior tibial nerve stimulation
  Arms: Electrical Stimulation
Other: Traditional treatment — Conventional treatment through Kegal exercises and dietetic regulation where they had received bulky food including vegetables, fruits bran and cereals. Fast foods, spicy drinks and caffeine should be limited in child's diet. Local hygiene and zinc oxide application to the perianal skin were advised to prevent skin excoriation.
  Other Names: Exercises
  Arms: Control group

SUMMARY:
Fecal incontinence is one of the most psychological frustrating problems. It occurs in children due to many causes. There is a wide range of non-invasive therapeutic approaches like Kegel exercise, Biofeedback, and posterior tibial nerve stimulation. However, up till now, there are no established guidelines for treatment.

the objective of this study is to evaluate and compare the early effect of Biofeedback therapy versus bilateral transcutaneous posterior tibial nerve stimulation (TPNS) as non-invasive methods in the treatment of functional non-retentive fecal incontinence (FNRFI) in children.

DETAILED DESCRIPTION:
Functional non-retentive fecal incontinence (FNRFI) requires prolonged treatment with a wide range of non-invasive therapeutic approaches like Kegel exercise, Biofeedback, and posterior tibial nerve stimulation (PTNS). However, up till now, there are no established guidelines for treatment.1 The aim of this study is to evaluate and compare the early effect of Biofeedback therapy versus bilateral transcutaneous posterior tibial nerve stimulation (TPTNS) as non-invasive methods in the treatment of (FNRFI) in children.

Methodology: The current prospective randomized controlled study included 93 children with FNRFI who were randomly divided and allocated into three groups. Group A treated by conventional methods through dietetic regulation and Kegal exercises. Group B treated by biofeedback therapy while group C received bilateral (TPTNS). Initial manometric findings including resting pressure, squeeze pressure, 1st sensation, 1st urge, and intense urge were recorded and repeated after 3 and 6 months together with incontinence score recorded in using St' Mark's (Varizey) with the primary endpoint of improvement of the incontinence score more than 50%.

ELIGIBILITY:
Inclusion Criteria:

* FecaI incontinence
* Normal defecation frequency,
* Normal bowel habits and
* Normal stool consistency

Exclusion Criteria:

* Children who are not cooperative,
* Children with traumatic sphincter injury,
* Children with fecal impaction,
* Children with spinal diseases causing incontinence,
* Children with anorectal malformation,

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Incontinence score using St' Mark's (Vaiszey) | 3 months after intervention
  Questionnaire ranging from zero (indicating complete continence) to 24 (indicating total incontinence).
incontinence score using St' Mark's (Vaiszey) | 6 months after intervention
  Questionnaire ranging from zero (indicating complete continence) to 24 (indicating total incontinence).

SECONDARY OUTCOMES:
Resting pressure (mm hg) | 3 months after intervention
  Pressure during relaxation of the anal sphincter
Resting pressure (mm hg) | 6 months after intervention
  Pressure during relaxation of the anal sphincter
Squeeze pressure (mm hg) | 3 months after intervention
  Pressure during contraction of the anal sphincter
Squeeze pressure (mm hg) | 6 months after intervention
  Pressure during contraction of the anal sphincter
First sensation (volume of the balloon by cm water) | 3 months after intervention
  First sensation of the stool in the rectum
First sensation (volume of the balloon by cm water) | 6 months after intervention
  First sensation of the stool in the rectum
First Urge(volume of the balloon by cm water) | 3 months after intervention
  The patient is trying to hold defecation and he can
First Urge(volume of the balloon by cm water) | 6 months after intervention
  The patient is trying to hold defecation and he can
Intense urge (volume of the balloon by cm water) | 3 months after intervention
  The Patent can no longer control the defecation
Intense urge (volume of the balloon by cm water) | 6 months after intervention
  the Patent can no longer control the defecation

CONTACTS AND LOCATIONS:
Overall Officials: Emad M Abdelrhman, PhD, Principal Investigator — Benha University
Locations (1):
- Banha University, Banhā, Banha, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After Publication, the investigators would like to share the data with authors interested in this topic
Supporting Information: Study Protocol
Time Frame: After Publication
Access Criteria: Not available now